CLINICAL TRIAL: NCT06167343
Title: Examining Anterior Cruciate Ligament Reconstruction With Quadriceps- vs. Semitendinosus Tendon Graft for Young Federated Male Football Players.
Brief Title: Comparison of Semitendinosus and Quadriceps Grafts for Anterior Cruciate Ligament Reconstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Hospital Vithas (Unknown)
Responsible Party: Principal Investigator, Maria Lopez-Garzon, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRUZADO23
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: ACL; ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semitendinosus tendon graft (Experimental): Surgical reconstruction of primary ACL rupture with autograft harvested from the semitendinosus tendon (ST).
  The ST graft is harvested through a 4-5 cm incision at the pes anserinus. The semitendinosus is identified and harvested. The tendon is prepared and folded to a four-stranded graft with a total diameter of 8-11 mm.
  The femoral tunnel is placed anatomically central in the native footprint of the ACL. The tibia tunnel is also placed anatomically; the center of the tunnel being medially between the eminential spines at the level of the posterior margin of the anterior horn of the lateral meniscus.
  The quadrupled ST graft is fixed proximally with the RIGIDLOOP® adjustable cortical system (DePuy Synthes) and distally with the RIGIDLOOP® XL adjustable cortical system.
  Interventions: Procedure: ACL reconstruction
- Quadriceps tendon graft (Experimental): Surgical reconstruction of primary ACL rupture with autograft harvested from the quadriceps tendon (QT) without bone block.
  The QT graft is harvested through a 4-5 cm incision at the upper pole of the patella. A graft sized 10-12 mm in with and app. 6 mm in depth is harvested from the middle part of the tendon.
  The femoral tunnel is placed anatomically central in the native footprint of the ACL. The tibia tunnel is also placed anatomically; the center of the tunnel being medially between the eminential spines at the level of the posterior margin of the anterior horn of the lateral meniscus.
  The QT graft is fixed proximally with the RIGIDLOOP® adjustable cortical system (DePuy Synthes) and distally with the RIGIDLOOP® XL adjustable cortical system
  Interventions: Procedure: ACL reconstruction

INTERVENTIONS:
Procedure: ACL reconstruction — In addition to surgical reconstruction, any structures that may have been injured concomitantly (meniscus, other ligament) will be repaired in the same surgery.

SUMMARY:
To investigate the differences between the two methods for reconstruction of the anterior cruciate ligament (ACL), to support the development of the best method for young federated male football players. After surgery with quadricipital tendon graft or semitendinosus tendon graft, a two-year follow-up and the rate of return to sport are proposed.

DETAILED DESCRIPTION:
The anterior cruciate ligament is one of the most common traumatic injuries in football, and surgery is proposed to restore knee stability. However, following surgery, few studies have focused on functional recovery of the knee with a wide arsenal of physical tests. Therefore, this study aims to study the efficacy for young football players of two types of grafts based on the most common tendons, the quadricipital and the semitendinosus (without the semimembranosus). Follow-ups will be performed at three months, six months, one year and two years after reconstruction. The variables measured will be isokinetic strength of flexors and extensors, unipodal jump test, self-perceived function, pain and tendon architecture with ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed anterior cruciate ligament rupture by MRI.
* Prognosis of anterior cruciate ligament reconstruction surgery.
* Be a registered or recreational football player.

Exclusion Criteria:

* Previous knee surgery.
* Having articular cartilage lesions of Outerbridge grade greater than III-IV.

Ages: 14 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Lower limb strength | Participants will be followed over 24 months
  assessed by an isokinetic test with an isokinetic dynamometer (HUMAC NORM)
Horizontal hop test | Participants will be followed over 24 months
  assessed by horizontal jump with one leg and hands on the waist, measured with a centimetric tape (three jumping opportunities)

SECONDARY OUTCOMES:
Self-reported functionality | Participants will be followed over 24 months
  assessed by Tegner Lysholm Knee Scoring Scale and Modified Cincinnati Rating System Questionnaire (Spanish version)
Knee pain | Participants will be followed over 24 months
  assessed by Visual Analogue Scale (VAS) for knee pain. The subjective perception of pain from 0 to 10 will be registered. Higher scores mean a worse outcome.
Pressure pain threshold | Participants will be followed over 24 months
  Using a digital algometer in epicondyle, vastus lateralis, vastus medialis and quadricipitalis tendon, patellar tendon, and insertion of the semitendinous tendon
Tendon ultrasound | Participants will be followed over 24 months
  it will monitor the morphology of the tendon and their surgical gap using ultrasound (Samsung HM70A echograph and Samsung Phased Array PE2-4 probe)
Perimeters | Participants will be followed over 24 months
  measured with the volume of both legs (injured and uninjured) using the mid-thigh circumference.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Granada, Granada, Spain